CLINICAL TRIAL: NCT00633854
Title: High-frequency-ultrasound Annular Arrays for Small Animal and Ophthalmic Imaging
Brief Title: High-frequency-ultrasound Annular Arrays for Ophthalmic Imaging
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Riverside Research Institute (Other)
Responsible Party: Ronald H. Silverman, PhD, Weill Cornell Medical College
Other Study IDs: EB008606
Record Dates: First submitted 2008-03-04; First posted 2008-03-12 (Estimated); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Posterior Vitreous Detachment
Keywords: annular array ultrasound; ophthalmic ultrasound; posterior vitreous detachment (PVD)
MeSH Terms: conditions — Vitreous Detachment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: 30 volunteer subjects who are age 60 and older
  Interventions: Procedure: Ultrasound examination

INTERVENTIONS:
Procedure: Ultrasound examination — Immersion Ultrasound Exam: In the immersion technique, the patient lies down on the examination table. A steridrape with a central aperture is used to form a water-tight seal around the eye. After installation of 2 drops of 0.5% proparacaine HCl, a wire lid speculum is used to hold the patient's lids open. Warm 0.9% sterile saline solution is then used to create a waterbath about 1/2 inch deep to provide acoustic coupling between the transducer and the eye. The transducer (either the 10- and 20-MHz sector scan probe or the annular array) is placed in the waterbath, but does not touch the eye.

SUMMARY:
The objective of this research is to improve the care of ocular disease and disorders, in particular the changes in the eye associated with diabetes, by providing clinicians with dramatically improved ultrasonic images of the entire eye. The research combines advanced high-frequency, high-resolution ultrasonic annular arrays transducers with new processing techniques designed to overcome several limits that have been reached with conventional high-frequency ultrasound systems. We propose that diagnosis of eye diseases using annular arrays can be more effective than the conventional ultrasound images by at least 50%; i.e., that for every 2 posterior vitreous detachments detected conventionally, 3 will be detected with the annular arrays.

DETAILED DESCRIPTION:
In this study, we will deploy annular-array systems and assess their experimental and clinical utility for ophthalmic imaging. We hypothesize that a 20-MHz annular array will detect posterior vitreous detachment (PVD) more reliably than a conventional single element ultrasound system. Clinically, we will test the hypothesis that 20-MHz annular arrays improve detection of PVD, an important risk factor for disease progression in diabetic retinopathy. Diabetic retinopathy is the leading cause of blindness in the working population (25 to 65 years) and the third major cause of legal blindness in the U.S.

We propose to carry out a study of 30 human subjects, aged 60 years or above, in whom PVD is likely to be present as a consequence of normal aging. The study will compare the ability to detect PVD using a commercial ophthalmic ultrasound system equipped with 10- and 20-MHz sector scan probes (Cinescan A/B-S, Quantel Medical), and OCT (OCT/SLO, Ophthalmic Technologies, Inc.), and the 20-MHz annular array. The annular array will be used with synthetic focusing and simulated single-element mode. The end point will be the fraction of eyes in which the PVD is visualized with each technique. This comparison is designed to demonstrate the improvement in our ability to visualize this pathologic entity using the advanced signal processing modes to be explored in this study. PVD can represent a risk factor for retinal detachment and retinal neovascularization in diabetics and localization of vitreoretinal traction points may be crucial for management. The present study, however, is limited to visualization of PVD in older normal subjects, about 75% of which would be expected to have PVD present. Thus, our aim is purely to develop an improved imaging modality rather than demonstrating its clinical efficacy in management of diabetic retinopathy or other ocular diseases.

The imaging technologies that we are developing could potentially result in patents or other intellectual property, which would be managed by the Cornell Research Foundation and Riverside Research Institute. This is alluded to in the consent form for the sake of completeness.

ELIGIBILITY:
Inclusion Criteria:

* Subjects should be age 60 or older with possible posterior vitreous detachment in the back of the eye.

Exclusion Criteria:

* none

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Ophthalmology practice
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2008-02; Primary Completion 2010-04-30 (Actual); Study Completion 2010-04-30 (Actual)

PRIMARY OUTCOMES:
detection of PVD in the posterior pole | outcome measured at time of examination

CONTACTS AND LOCATIONS:
Overall Officials: Ronald H Silverman, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

REFERENCES:
- [Background] Silverman RH, Ketterling JA, Mamou J, Coleman DJ. Improved high-resolution ultrasonic imaging of the eye. Arch Ophthalmol. 2008 Jan;126(1):94-7. doi: 10.1001/archopht.126.1.94. PMID 18195224
- [Background] Silverman RH, Ketterling JA, Coleman DJ. High-frequency ultrasonic imaging of the anterior segment using an annular array transducer. Ophthalmology. 2007 Apr;114(4):816-22. doi: 10.1016/j.ophtha.2006.07.050. Epub 2006 Nov 30. PMID 17141314